CLINICAL TRIAL: NCT02157233
Title: Post-exercise Food Intake Regulation in a Hot Environment
Acronym: APPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the French West Indies and French Guiana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 13/N/01
Record Dates: First submitted 2014-06-02; First posted 2014-06-05 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Healthy and Physically Active Young Men
MeSH Terms: interventions — RE1-silencing transcription factor; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hot environment (Experimental): Subjects will perform the intervention in a hot environment (33°C)
  Interventions: Behavioral: Rest; Behavioral: Exercise
- Neutral environment (Sham Comparator): Subjects will perform the intervention in a neutral environment (22°C)
  Interventions: Behavioral: Rest; Behavioral: Exercise

INTERVENTIONS:
Behavioral: Rest
Behavioral: Exercise

SUMMARY:
The potential of physical activity and other non-medicinal methods for the care and prevention of metabolic and cardiovascular disorders has been insufficiently used. There is a potential influence of environmental heat in energetic balance regulation. However, the existing knowledge is insufficient to optimize physical activity programs based on the impact of exercise on energy intake regulation in hot climates. The aim of the present study is to define the major physiological determinants of short-term food intake regulation in young active and healthy men, when exposed to different levels of metabolic activity and environmental temperatures. We will thus explore the biological mechanisms related to post-exercise relative energy intake. Post-rest and post-exercise energetic compensation will be analysed in these different environmental conditions, with a special focus on the effect of the birth weight. This study should open interesting ways to define adequate nutritional and exercising programs in hot environments.

ELIGIBILITY:
Inclusion Criteria:

* healthy and physically active men aged 18-30 years

Exclusion Criteria:

* any physical or medical problem liable to limit the subjects' ability to perform the exercise testing in safe conditions,
* ear troubles

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-10; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Relative post-exercise and post-rest energy intake | 11 months

SECONDARY OUTCOMES:
Appetite hormones | 13 months
  insulin, CCK, leptin, ghrelin, pancreatic peptide
Heart rate variability | 11 months
Tympanic temperature | 11 months
Peak exercise capacity | 11 months
Appetite visual analogic scale | 11 months
metabolic markers | 13 months
  glucose, lipid profile, cortisol
vascular biomarkers | 13 months
  usCRP, inflammatory markers, hemorheological markers
comfort visual scale | 11 months

CONTACTS AND LOCATIONS:
Locations (1):
- CREPS, Les Abymes, Guadeloupe, France

REFERENCES:
- [Derived] Faure C, Charlot K, Henri S, Hardy-Dessources MD, Hue O, Antoine-Jonville S. Effect of heat exposure and exercise on food intake regulation: A randomized crossover study in young healthy men. Metabolism. 2016 Oct;65(10):1541-9. doi: 10.1016/j.metabol.2016.07.004. Epub 2016 Jul 11. PMID 27621189